CLINICAL TRIAL: NCT01863368
Title: Clinical Evaluation of Systane® ULTRA Compared to OPTIVE® in Ocular Surface Staining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-12-040
Record Dates: First submitted 2013-05-23; First posted 2013-05-27 (Estimated); Results first posted 2015-07-10 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Dry Eye Syndrome
Keywords: Dry eye syndrome; Systane Ultra; Optive; Ocular Surface Staining; OSDI; Eye drops
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane Ultra (Experimental): Systane® ULTRA lubricant eyedrops, 1 drop in each eye 4 times a day for 35 days (Phase I), followed by 55 days additional use as needed (Phase II).
  Interventions: Other: Preservative-free saline solution eyedrops; Other: Systane® ULTRA lubricant eyedrops
- Optive (Active Comparator): OPTIVE® lubricating eyedrops, 1 drop in each eye 4 times a day for 35 days (Phase I), followed by 55 days additional use as needed (Phase II).
  Interventions: Other: Preservative-free saline solution eyedrops; Other: OPTIVE® lubricating eyedrops

INTERVENTIONS:
Other: Preservative-free saline solution eyedrops — 1 drop in each eye, 4 times a day, for up to two weeks as washout prior to Phase I and Phase II.
Other: Systane® ULTRA lubricant eyedrops
  Arms: Systane Ultra
Other: OPTIVE® lubricating eyedrops
  Arms: Optive

SUMMARY:
The purpose of this study is to compare Systane® ULTRA lubricant eye drops to OPTIVE® lubricating eye drops for ocular surface staining within dry eye subjects and to evaluate the safety of Systane® ULTRA after 3 months of use.

DETAILED DESCRIPTION:
Following a 2-week washout phase with saline eye drops, subjects were randomized to receive either Systane® ULTRA or OPTIVE® for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to attend all study visits.
* Diagnosis of dry eye, as specified in protocol.
* Uses artificial tears, as specified in protocol.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Poor visual acuity, as specified in protocol.
* Women of childbearing potential who are pregnant, lactating, or not using adequate birth control, as specified in protocol.
* Any hypersensitivity or allergy to the investigational products or ingredients.
* Any eye disorder, ocular surgery, medication, medical condition, or systemic disease, as specified in protocol.
* Contact lens use within 2 weeks of Screening Visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Burmaster, Study Director — Alcon Research

REFERENCES:
- [Derived] Labetoulle M, Messmer EM, Pisella PJ, Ogundele A, Baudouin C. Safety and efficacy of a hydroxypropyl guar/polyethylene glycol/propylene glycol-based lubricant eye-drop in patients with dry eye. Br J Ophthalmol. 2017 Apr;101(4):487-492. doi: 10.1136/bjophthalmol-2016-308608. Epub 2016 Jul 15. PMID 27422973

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 13 study centers located in France and 3 study centers located in Germany.
Pre-assignment Details: Of the 105 enrolled, 11 subjects were exited prior to randomization: 9 screen failures, 1 adverse event, and 1 lost to follow-up. This reporting group includes all randomized subjects (94).
Groups:
- Systane Ultra: Lubricant eyedrops, 1 drop in each eye 4 times a day for 35 days (Phase I), followed by 55 days additional use as needed (Phase II).
- Optive: Lubricating eyedrops, 1 drop in each eye 4 times a day for 35 days (Phase I), followed by 55 days additional use as needed (Phase II).
Period: Phase I, Day 0 to Day 35
Arm/Group | Systane Ultra | Optive
Started | 46 | 48
Treated | 46 | 47
Completed | 43 | 41
Not Completed | 3 | 7
Not completed — Adverse Event | 2 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by subject prior to treatment | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Period: Phase II, Day 35 to Day 90
Arm/Group | Systane Ultra | Optive
Started | 43 | 41
Completed | 41 | 41
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis group includes all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Systane Ultra | Optive | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (13.1) | 65.2 (14.3) | 64.4 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 7 | 8 | 15
Mean Total Ocular Surface Staining (TOSS) Score [Mean (Standard Deviation); unit: units on a scale] — The TOSS score is a composite score of corneal fluorescein staining, nasal conjunctival lissamine green staining, and temporal conjunctival lissamine green staining, each scored on a 0-5 Likert scale (0=absent, 5=severe). TOSS scores can range from 0 to 15. One eye (study eye) contributed to the analysis. Here, the analysis group includes all randomized subjects with data at visit (46,47 respectively, for a total of 93).
  units on a scale | 5.5 (1.9) | 5.5 (1.7) | 5.5 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Ocular Surface Staining (TOSS) Score at Day 35 (Phase I)
Description: The TOSS score is a composite score of corneal fluorescein staining, nasal conjunctival lissamine green staining, and temporal conjunctival lissamine green staining, each scored on a 0-5 Likert scale (0=absent, 5=severe). TOSS scores can range from 0 to 15. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Day 35
Population: This analysis group includes all randomized subjects with data at visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Systane Ultra | Optive
Number analyzed (Participants) | 43 | 41
units on a scale | -2.2 (2.3) | -1.7 (2.4)

2. Secondary Outcome: Mean Ocular Surface Disease Index (OSDI) Score at Day 35 (Phase I)
Description: The OSDI is a 12-item, quality of life questionnaire that evaluates symptoms based on 3 modules (type of discomfort, environmental triggers, and tasking) on a 0-4 Likert scale (0=None of the time, 4=All of the time). A resultant overall 0-100 score was calculated, where 0=No disability and 100=Complete disability. Both eyes contributed to the analysis.
Time Frame: Day 35
Population: This analysis group includes all subjects with data at visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Systane Ultra | Optive
Number analyzed (Participants) | 43 | 41
units on a scale | 31.0 (18.3) | 35.4 (17.1)

3. Secondary Outcome: Mean Impact of Dry Eye on Everyday Life (IDEEL) Treatment Effectiveness Score at Day 35 (Phase I)
Description: The IDEEL is a 10-item, patient-reported questionnaire used to measure treatment satisfaction. The subject answered 4 questions pertaining to treatment effectiveness scored on a 0-4 Likert-type scale, where 0=None of the time, 1=A little of the time, 2=Some of the time, 3=Most of the time, and 4=All of the time. The IDEEL score for treatment effectiveness was calculated based upon the mean value of the 4 questions multiplied by 25, for a resultant overall score of 0-100, where 0=Complete disability and 100=No disability. Both eyes contributed to the analysis.
Time Frame: Day 35
Population: This analysis group includes all subjects with data at visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Systane Ultra | Optive
Number analyzed (Participants) | 43 | 41
units on a scale | 62.2 (27.3) | 55.7 (29.4)

4. Secondary Outcome: Mean Impact of Dry Eye on Everyday Life (IDEEL) Treatment Inconvenience Score at Day 35 (Phase I)
Description: The IDEEL is a 10-item, patient-reported questionnaire used to measure treatment satisfaction. The subject answered 4 questions pertaining to treatment inconvenience scored on a 0-4 Likert-type scale, where 0=All of the time, 1=Most of the time, 2=Some of the time, 3=A little of the time, and 4=None of the time. The IDEEL score for treatment inconvenience was calculated based upon the mean value of the 4 questions multiplied by 25, for a resultant overall score of 0-100, where 0=Complete disability and 100=No disability. Both eyes contributed to the analysis.
Time Frame: Day 35
Population: This analysis group includes all subjects with data at visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Systane Ultra | Optive
Number analyzed (Participants) | 43 | 41
units on a scale | 69.5 (15.8) | 67.1 (23.6)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (Sep 2013 - Jun 2014). AEs are reported as pre-treatment and treatment-emergent. One subject was randomized to Optive, but was never exposed to product.
Description: An AE was defined as any untoward medical occurrence in a subject who was administered an investigational product regardless of whether or not the event had a causal relationship with the product. AEs were obtained as solicited and spontaneous comments from the study subjects, and as observations by the Investigator, as outlined in the protocol.
Groups:
- Pre-treatment: All subjects who consented to participate in the study prior to exposure to investigational product
- Systane Ultra: All subjects who were exposed to Systane Ultra or run-in therapy
- Optive: All subjects who were exposed to Optive or run-in therapy
Arm/Group | Pre-treatment | Systane Ultra | Optive
Serious Adverse Events (participants affected / at risk) | 1/105 | 1/46 | 0/47
Other Adverse Events (participants affected / at risk) | 1/105 | 2/46 | 3/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-treatment (N=105) | Systane Ultra (N=46) | Optive (N=47)
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-treatment (N=105) | Systane Ultra (N=46) | Optive (N=47)
Eye irritation (Eye disorders) | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.